CLINICAL TRIAL: NCT06106945
Title: A Modular Phase I/II, Open-label, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Lmmunogenicity, Pharmacodynamics, and Preliminary Efficacy of AZD0305 as Monotherapy or in Combination With Anticancer Agent(s) in Participants With Relapsed or Refractory Multiple Myeloma
Brief Title: AZD0305 as Monotherapy or in Combination With Anticancer Agents in Participants With Relapsed/Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7230C00001; 2023-508590-89-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-10-11; First posted 2023-10-30 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: GPRC5D; ADC; AZD0305; Relapsed Refractory Multiple Myeloma; RRMM; MMAE
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: This protocol has a modular design, with the potential for future treatment arms, study parts, or modules to be added via protocol amendments. Module 1 will include Phase Ia (Dose escalation), and Phase Ib (Dose expansion/optimization).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD0305 monotherapy (Experimental): Module 1:
  Phase Ia: Dose Escalation Phase Ib: Dose Expansion/Optimization AZD0305 will be prescribed at specified dose levels.
  Interventions: Drug: AZD0305

INTERVENTIONS:
Drug: AZD0305 — AZD0305

SUMMARY:
This is a Phase I/II, modular, open-label, multicenter, dose escalation, and dose expansion/optimization study to evaluate the safety, tolerability, PK, immunogenicity, pharmacodynamics, and preliminary efficacy of AZD0305 in participants with RRMM.

DETAILED DESCRIPTION:
This is a Phase I/II, modular, open-label, multicenter, dose escalation, and dose expansion/optimization study to evaluate the safety, tolerability, PK, immunogenicity, pharmacodynamics, and preliminary efficacy of AZD0305 in participants with RRMM. This study will follow a modular protocol design evaluating AZD0305 as monotherapy and in combination with other anticancer agents.

The study includes dose escalation and dose expansion phases. This study will enroll subjects with RRMM who received at least 3 prior lines of treatment including at least one proteasome inhibitor (PI), one immunomodulator (IMiD), and an anti-CD38 antibody.

ELIGIBILITY:
Principal Inclusion Criteria:

* Participants must be at least 18 years of age or the legal age of consent in the jurisdiction in which the study is taking place.
* Eastern Cooperative Oncology group (ECOG) performance status of ≤ 2.
* Documentation of Multiple Myeloma (MM) as defined by International Myeloma Working Group (IMWG) Diagnostic Criteria for Multiple Myeloma. Site should ensure that Multiple Myeloma diagnosis is confirmed in accordance with the IMWG Diagnostic Criteria.
* Participants must have one or more of the following measurable disease criteria:

  1. Serum M-protein level ≥ 0.5 g/dL.
  2. Urine M-protein level ≥ 200 mg/24h.
  3. Serum immunoglobulin free light chain ≥ 10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio.
* Adequate organ and bone marrow function assessment at screening according to the hematological, hepatic, and renal parameters listed in the CSP.
* Participants must have received at least 3 prior lines of treatment which include a proteasome inhibitor (e.g., bortezomib), an immunomodulator (e.g., lenalidomide), and an anti-CD38 antibody (e.g., daratumumab).

Principal Exclusion Criteria:

* Participants exhibiting clinical signs of central nervous system involvement of MM.
* Participants with known COPD, or previous history of ILD.
* Participants with known moderate or severe persistent asthma within the past 5 years, or uncontrolled asthma of any classification.
* Participants who have severe cardiovascular disease which is not adequately controlled.
* Participants who have a history of immunodeficiency disease.
* Participants with peripheral neuropathy ≥ Grade 2.
* Primary refractory MM.
* Participants who have previously received anti-GPRC5D or MMAE-containing treatment.
* Participants who have previously received allogenic stem cell transplant, or participant has received autologous stem cell transplant within 3 months before the first dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2027-08-16 (Estimated); Study Completion 2027-08-16 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicity (DLT), as defined in the protocol (Phase Ia dose escalation only) | From first dose of study treatment until the end of Cycle 1
  A DLT is defined as any toxicity that occurs from the first dose of study treatment up to and including the planned end of Cycle 1 (the DLT assessment period) that is assessed as unrelated to the disease or disease-related processes under investigation and which includes, any death not clearly due to the underlying disease or extraneous causes, pre-defined haematological and non-haematological toxicities
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From time of Informed consent to 30 days post end of treatment
  Number of patients with adverse events and serious adverse events by system organ class and preferred term

SECONDARY OUTCOMES:
Phase Ia: Objective Response Rate (ORR) | From first dose of AZD0305 to progressive disease or Initiation of subsequent MM therapy (approximately 2 years)
  The percentage of patients with a confirmed investigator assessed sCR, CR, VGPR or PR according to IMWG criteria
Phase Ia: Duration of response (DoR) | From the first documented response to confirmed progressive disease or death (approximately 2 years)
  The time from the date of first response until date of disease progression or death in the absence of disease progression
Phase Ia: Progression free Survival (PFS) | From first dose of AZD0305 to progressive disease or death in the absence of disease progression (approximately 2 years)
  The time from first dose until IMWG defined disease progression or death
Phase Ia: Overall Survival (OS) | From first dose of AZD0305 to death (approximately 2 years)
  The time from the date of the first dose of study treatment until death due to any cause
Phase Ia: Pharmacokinetics of AZD0305: Area Under the concentration-time curve (AUC) | From the first dose of study intervention, at predefined intervals throughout the administration of AZD0305 (approximately 2 years)
  Area under the plasma concentration-time curve
Phase Ia: Pharmacokinetics of AZD0305: Maximum plasma concentration of the study drug (Cmax) | From the first dose of study intervention, at predefined intervals throughout the administration of AZD0305 (approximately 2 years)
  Maximum observed plasma concentration of the study drug
Phase Ia: Pharmacokinetics of AZD0305: Time to maximum plasma concentration of the study drug (tmax) | From the first dose of study intervention, at predefined intervals throughout the administration of AZD0305 (approximately 2 years)
  Time to maximum observed plasma concentration of the study drug
Phase Ia: Pharmacokinetics of AZD0305: Clearance | From the first dose of study intervention, at predefined intervals throughout the administration of AZD0305 (approximately 2 years)
  A pharmacokinetic measurement of the volume of plasma from which the study drug is completely removed per unit time
Phase Ia: Pharmacokinetics of AZD0305: Terminal elimination half-life (t 1/2) | From the first dose of study intervention, at predefined intervals throughout the administration of AZD0305 (approximately 2 years)
  Terminal elimination half-life
Phase Ia: Immunogenicity of AZD0305 | From the first dose of study intervention, at predefined intervals throughout the administration of AZD0305 (approximately 2 years)
  The number and percentage of participants who develop ADAs
Phase Ib: Objective Response Rate (ORR) | From randomization to progressive disease or Initiation of subsequent MM therapy (approximately 2 years)
  The percentage of patients with a confirmed investigator assessed sCR, CR, VGPR or PR according to IMWG criteria
Phase Ib: Duration of response (DoR) | From randomization to confirmed progressive disease or death (approximately 2 years)
  The time from date of first response until date of disease progression or death in the absence of disease progression
Phase Ib: Progression free Survival (PFS) | From randomization to progressive disease or death in the absence of disease progression (approximately 2 years)
  The time from randomization until IMWG defined disease progression or death
Phase Ib: Overall Survival (OS) | From randomization to death (approximately 2 years)
  The time from randomization until death due to any cause
Phase Ib: Pharmacokinetics of AZD0305: Area Under the concentration-time curve (AUC) | From randomization, at predefined intervals throughout the administration of AZD0305 (approximately 2 years)
  Area under the plasma concentration-time curve
Phase Ib: Pharmacokinetics of AZD0305: Maximum plasma concentration of the study drug (Cmax) | From randomization, at predefined intervals throughout the administration of AZD0305 (approximately 2 years)
  Maximum observed plasma concentration of the study drug
Phase Ib: Pharmacokinetics of AZD0305: Time to maximum plasma concentration of the study drug (tmax) | From randomization, at predefined intervals throughout the administration of AZD0305 (approximately 2 years)
  Time to maximum observed plasma concentration of the study drug
Phase Ib: Pharmacokinetics of AZD0305: Clearance | From randomization, at predefined intervals throughout the administration of AZD0305 (approximately 2 years
  A pharmacokinetic measurement of the volume of plasma from which the study drug is completely removed per unit time
Phase Ib: Pharmacokinetics of AZD0305: Terminal elimination half-life (t 1/2) | From randomization, at predefined intervals throughout the administration of AZD0305 (approximately 2 years)
  Terminal elimination half-life
Phase Ib: Immunogenicity of AZD0305 | From randomization, at predefined intervals throughout the administration of AZD0305 (approximately 2 years)
  The number and percentage of participants who develop ADAs

CONTACTS AND LOCATIONS:
Locations (35):
- United States (9):
  - Research Site, Duarte, California
  - Research Site, Irvine, California
  - Research Site, Atlanta, Georgia
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Fairfax, Virginia
- Australia (2):
  - Research Site, Melbourne
  - Research Site, Nedlands
- Canada (4):
  - Research Site, Hamilton, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Nova Scotia
- China (4):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Guangzhou
  - Research Site, Shenyang
- France (2):
  - Research Site, Lille
  - Research Site, Nantes
- Germany (8):
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Lübeck
  - Research Site, Nuremberg
  - Research Site, Tübingen
  - Research Site, Würzburg
- Japan (3):
  - Research Site, Kashiwa
  - Research Site, Nagoya
  - Research Site, Yamagata
- Spain (3):
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home